CLINICAL TRIAL: NCT06818344
Title: Sensory Modulation in Children With Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor Dr., Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-7
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy; Sensory Modulation Disorder
Keywords: epilepsy; sensory modulation; child
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: Children diagnosed with epilepsy constitute the "case group." Sensory modulation assessments will be conducted for the children in this group.
- Control group: The control group consists of healthy children. The same assessment will be applied to this group as well.

SUMMARY:
Epilepsy is a neurological condition that can impact cognitive, motor, and behavioral skills, often leading to sensory modulation disorders (SMDs) in children. These disorders impair sensory processing, affecting daily functioning and quality of life. This study aims to explore the sensory profiles of children with epilepsy and identify sensory modulation disorders.

The study will include 34 participants: 17 children with epilepsy and 17 healthy controls, aged 3-10 years. Inclusion criteria include at least one seizure in the past year, a diagnosis of epilepsy, and voluntary participation. Children with comorbid conditions such as cerebral palsy, autism, genetic disorders, or other neurological conditions will be excluded.

Data on demographics and epilepsy-related characteristics will be gathered from families. Sensory modulation will be assessed using the Sensory Profile, a 125-item Likert-type questionnaire completed by parents. It evaluates sensory processing across three categories: sensory processing, sensory modulation, and behavioral-emotional responses. Results will classify children as "Typical Performance," "Probable Difference," or "Definite Difference." Data will be analyzed using IBM SPSS 26.0 and R Software. The Shapiro-Wilk test will assess normality, followed by an Independent Samples t-test or Mann-Whitney U Test depending on data distribution. The Chi-Square test will be used for categorical variables.

This study aims to identify the prevalence and types of sensory modulation disorders in children with epilepsy. While previous studies suggest sensory processing issues in children with epilepsy, they often involve small samples. By using a larger sample, this research will provide stronger insights into the sensory profiles of children with epilepsy. The findings may contribute to earlier diagnosis and intervention strategies.

Future research should involve larger samples and longitudinal designs to investigate long-term effects and therapeutic approaches for sensory modulation disorders, ultimately improving the quality of life for children with epilepsy.

DETAILED DESCRIPTION:
Epilepsy is a transient condition resulting from abnormal hyperactivity of neurons or desynchronized neuronal circuits in the brain, as defined by the International League Against Epilepsy. It is one of the most common chronic diseases of childhood, affecting approximately 0.5-1% of children worldwide. According to relevant literature, an estimated 10.5 million children under the age of 15 are currently being monitored with an active epilepsy diagnosis. Epilepsy is classified based on clinical characteristics, including seizure type, age of onset, cognitive and developmental history, presence of neurological symptoms, family history, electroencephalography (EEG) findings, seizure triggers, sleep-related seizure frequency, and prognosis. Seizures in children with epilepsy have profound negative effects on social, psychological, and physical health, leading to impairments in cognitive functions. Various studies have demonstrated that children with epilepsy exhibit potential deficits in intelligence, memory, learning, attention, motor skills, and behavioral abilities. Additionally, deficits in executive functions and motor coordination have been reported, along with difficulties in developing appropriate skills in response to environmental demands.

In addition to epilepsy, sensory processing disorders (SPDs) significantly affect children's ability to process, regulate, and interpret sensory information from their environment. These disorders influence cognitive, motor, behavioral, and emotional responses. SPDs often result in impairments in neuropsychomotor development. Children experiencing these difficulties may exhibit behavioral problems, sleep disturbances, social interaction challenges, and aggression. Furthermore, heightened emotional responses and excessive crying are frequently observed behavioral characteristics in these children. Self-regulation, learning, functional behaviors, daily living skills, movement organization, and school performance can also be negatively impacted by sensory processing disorders. SPDs are generally classified into three main categories: sensory modulation disorder, sensory-based motor disorder, and sensory discrimination disorder.

According to Dunn's sensory processing framework, individuals' responses to sensory stimuli vary based on their neurological thresholds and the type of response they exhibit to stimuli. Dunn suggests a continuous interaction between sensory input and individual responses, which may lead to atypical behaviors if adaptation to stimuli is inadequate. She categorizes responses into passive and active self-regulation strategies. Passive self-regulation involves experiencing stimuli without altering them, whereas active self-regulation involves controlling and modifying sensory input. Based on this model, four distinct sensory profiles are identified: low registration, sensory seeking, sensory sensitivity, and sensory avoidance. Low registration refers to individuals with a high neurological threshold, meaning they fail to notice or respond slowly to sensory stimuli. Sensory seeking describes individuals with a high sensory threshold who actively seek intense stimuli, such as strong smells, loud noises, or bright lights. Sensory sensitivity refers to individuals with a low sensory threshold who perceive stimuli but do not actively respond to them. Sensory avoidance, on the other hand, involves individuals with a low sensory threshold who develop active strategies to avoid distressing stimuli.

Sensory modulation disorders (SMDs) involve difficulties in detecting, regulating, and interpreting sensory stimuli, as well as disruptions in the responses given to sensory input. In the literature, sensory modulation disorders are categorized into three main groups: sensory over-responsivity, sensory under-responsivity, and sensory seeking. These disorders can lead to behavioral issues due to the inability to regulate responses to sensory stimuli from the environment.

Studies on children with epilepsy have often been conducted with small sample sizes and have focused on specific types of epilepsy, frequently using only the short form of sensory profiles. As a result, findings from these studies cannot be generalized to all types of epilepsy. Despite these limitations, existing research highlights the need for further studies on the prevalence and effects of sensory modulation disorders in children with epilepsy.

Objectives:

To assess sensory modulation in children with epilepsy. To investigate the sensory profiles of children with epilepsy. To compare sensory modulation across different types of epilepsy. To compare sensory modulation abilities between children with epilepsy and healthy peers.

This study aims to contribute to clinical practice and scientific research by providing comprehensive data on sensory modulation in children with epilepsy. By identifying sensory modulation disorders in a larger sample of children with epilepsy, this research seeks to enhance understanding and support the development of effective early diagnostic methods and interventions. Ultimately, this study aspires to fill gaps in the literature and promote interventions that improve the daily living skills and overall well-being of children with epilepsy.

This study is planned to include 17 children with epilepsy and 17 healthy children aged 3-10 years, whose families have agreed to participate. During the study period, children meeting the inclusion criteria will be evaluated. Participants will be selected based on voluntary participation and their compatibility with the inclusion criteria. General demographic information and detailed data regarding epilepsy-related characteristics will be collected. Families will be asked about the age of seizure onset, seizure frequency, medications used, comorbid conditions, and family history of psychiatric disorders. The presence of cerebellar pathology in participating children will be examined through a neurological assessment conducted by the neurologist involved in the study. Sensory modulation will be assessed using the Sensory Profile test, and the results of children with epilepsy and healthy children will be compared.

Sensory Profile

The Sensory Profile test will be used to assess the sensory processing status of the children included in our study. It was developed by Winnie Dunn. This test evaluates how children aged 3-10 process information received from their bodies and surroundings. It is a five-point Likert-type parent questionnaire consisting of 125 items. The Turkish version was developed by Kayihan et al. in 2015. Before starting the questionnaire, the child's name, date of birth, the respondent's identity and relationship to the child, the service provider, the institution, and the date of administration are recorded. The caregiver is instructed to mark the option that best describes how frequently the child exhibits the behaviors listed in the questionnaire and to provide answers for all parameters. If the caregiver has never observed a behavior or believes it does not apply to the child, they are instructed to mark an "X" for that item.

The questionnaire is divided into three main categories: Sensory Processing, Modulation, and Behavioral and Emotional Responses.

Sensory Processing: Includes subcategories such as auditory processing, visual processing, vestibular processing, tactile processing, multisensory processing, and oral sensory processing.

Modulation: Includes subcategories related to sensory processing in relation to endurance/tone, movement and body position, movement affecting activity levels, regulation of sensory input affecting emotional responses, and regulation of visual input affecting emotional responses and activity levels.

Behavioral and Emotional Responses: Includes subcategories related to emotional and social responses, behavioral outcomes of sensory processing, and threshold levels for response.

Each section is scored based on the frequency of behaviors using the following scale: Always (1), Frequently (2), Occasionally (3), Seldom (4), Never (5). The total score for each section is calculated, and children are classified into categories according to Dunn's Sensory Profile Scoring Interpretation: Definite Difference, Probable Difference, or Typical Performance.

Typical Performance: Indicates normal sensory processing development.

Definite Difference: Suggests the presence of sensory processing disorder.

Probable Difference: Suggests the possibility of sensory processing disorder and indicates the need for clinical evaluation.

The Sensory Processing section provides results related to auditory processing, visual processing, vestibular processing, tactile processing, multisensory processing, oral sensory processing, endurance and tone-related sensory processing, movement and body position regulation, movement affecting activity levels, sensory input regulation affecting emotional responses, regulation of visual input affecting emotional responses and activity levels, emotional and social responses, behavioral outcomes of sensory processing, and threshold levels for response.

The Modulation section provides results related to sensory seeking, emotional response, low endurance/tone, oral sensory sensitivity, inattentiveness/distractibility, poor registration, sensory sensitivity, sedentary behavior, and perceptual fine motor processing.

The Behavioral and Emotional Responses section provides results related to registration, exploration, sensitivity, and avoidance.

A literature review revealed no direct studies on sensory perception in the relevant population. However, studies in the literature suggest that sensory perception and sensory modulation yield similar outcomes. Therefore, a study measuring sensory modulation was considered. In this study, a large effect size (d = 1.31) was observed between patient and control groups. Based on this effect size, the required sample size was calculated for an independent samples t-test, considering a power of 90% and a 5% type I error rate. It was determined that at least 14 participants per group, totaling a minimum of 28 participants, would be required. Assuming a 20% dropout rate per group, the study aimed to include at least 34 participants, with 17 in each group. The sample size calculation was performed using G*Power 3.1.9.7.

For statistical analyses, IBM SPSS Statistics for Windows, version 26.0 (Armonk, NY: IBM), and R Statistical Software (v4.3.0; R Core Team, 2023) will be used. Descriptive statistics will be reported as mean and standard deviation or quartiles for numerical variables, and as frequency and percentage for categorical variables. Normality assumptions will be assessed using graphical methods (QQ plots, histograms, etc.) and hypothesis tests (Shapiro-Wilk test). For the comparison of numerical variables between two groups, an independent samples t-test will be conducted if assumptions are met, whereas the Mann-Whitney U test will be used if assumptions are violated. For categorical variables, chi-square test statistics (Pearson, Yates, Fisher's exact test, etc.) will be employed. Correlations between numerical variables will be analyzed using Pearson or Spearman correlation coefficients, depending on the assumption of normality. A significance level of p < 0.05 will be adopted.

ELIGIBILITY:
Inclusion Criteria:

Having had a seizure in the year prior to data collection Clinical diagnosis of epilepsy Aged between 3 and 10 years Willing to participate in the study

Exclusion Criteria:

Diagnosis of cerebral palsy Diagnosis of hydrocephalus Diagnosis of autism spectrum disorder Diagnosis of pervasive developmental disorder Diagnosis of learning disabilities Diagnosis of dyslexia Diagnosis of genetic disorders Diagnosis of metabolic disorders Diagnosis of neuromuscular diseases

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3-10 years diagnosed with epilepsy and healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sensory Profile | 1 year
  The Sensory Profile, developed by Winnie Dunn, is a 125-item Likert-type questionnaire used to assess how children aged 3-10 process sensory information from their bodies and environment. It is divided into three main sections: Sensory Processing, Modulation, and Behavioral and Emotional Responses. Sensory Processing includes subcategories such as auditory, visual, vestibular, tactile, multisensory, and oral processing. Modulation evaluates sensory processing related to endurance, movement, and body position, as well as the regulation of sensory inputs affecting emotional responses. Behavioral and Emotional Responses assess emotional, social responses, and behavioral consequences. Each section is scored based on frequency, and children are classified as having "typical performance," "probable difference," or "definite difference," based on the results. The test is widely used to evaluate sensory processing disorders in children.

CONTACTS AND LOCATIONS:
Overall Officials: Seda AYAZ TAS, PhD, Study Director — Abant Izzet Baysal University
Locations (1):
- Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Campen JS, Jansen FE, Kleinrensink NJ, Joels M, Braun KP, Bruining H. Sensory modulation disorders in childhood epilepsy. J Neurodev Disord. 2015;7:34. doi: 10.1186/s11689-015-9130-9. Epub 2015 Oct 23. PMID 26504494